CLINICAL TRIAL: NCT04527419
Title: Systematically Mediastinal Lymph Node Dissection or Not in Stage T1 Ground-glass Dominated Invasive Lung Adenocarcinoma: a Multi-center, Prospective Clinical Trial
Brief Title: SLND or Not in cT1 GGO Invasive Lung Adenocarcinoma (ECTOP-1009)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Haiquan Chen, Director, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SLNDILA
Record Dates: First submitted 2020-08-23; First posted 2020-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: invasive lung adenocarcinoma; systematically mediastinal lymph node dissection; ground-glass nodule
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Masking Description: Treatment groups will be open to both patients and surgeons.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- No mediastinal lymph node dissection group (Experimental): Mediastinal lymph node dissection will not be performed.
  Interventions: Procedure: No mediastinal lymph node dissection

INTERVENTIONS:
Procedure: No mediastinal lymph node dissection — No mediastinal lymph node dissection will be performed.

SUMMARY:
This is a study from Eastern Cooperative Thoracic Oncology Project, numbered as ECTOP-1009. Systematically mediastinal lymph node dissection or not in clinical stage T1 ground-glass dominated invasive lung adenocarcinoma: a multi-center, prospective clinical trial

DETAILED DESCRIPTION:
Following interim analysis of 302 patients revealed no lymph node metastasis in either study arm and 100% 2-year disease-free survival in both arms. The selective non-mediastinal lymph node dissection (non-SLND) arm had reduced complications (JCO 2025; doi:10.1200/JCO-25-00610). The study design has been amended to a single-arm prospective cohort. All enrolled patients meeting inclusion criteria will sign informed consent and receive non-SLND. The primary endpoint remains 3-year disease-free survival (DFS).

The sample size has been recalibrated to 545 patients based on historical control 3-year DFS of 96.6%, a stricter non-inferiority margin of 2.5%, 90% power, and the 1-sided alpha of 2.5%.

ELIGIBILITY:
Inclusion Criteria:

* Clinical stage T1N0M0 and planned curative surgery.
* A single lesion detected on computed tomography (CT) scan featured as ground glass nodule(GGO) and C/T ratio ≤0.5.
* Age 18 to 75.
* Patients who have signed the informed consent form.

Exclusion Criteria:

* Other than invasive adenocarcinoma by pathological analysis.
* Patients undergoing wedge resection but not meeting the specific conditions of a Consolidation/Tumor Ratio (CTR) ≤ 0.25 AND a maximum tumor diameter ≤ 2 cm, based on the oncological outcomes of the JCOG0804/WJOG4507L trial.
* Not complete resected or curative intent.
* Patients who have history of other malignant tumors.
* Patients who have history of thoracic surgery.
* Patients who have received radiation, chemotherapy or other treatments previously.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 545 (Estimated)
Dates: Start 2022-02-09 (Actual); Primary Completion 2026-07-21 (Estimated); Study Completion 2027-02-09 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 3 years after the surgery
  Disease-free survival means the period after surgery when no disease can be detected.

SECONDARY OUTCOMES:
Overall survival | 3 years after the surgery
  Overall survival means the period after surgery when a patient doesn't die directly from lung cancer or an unrelated cause.
Rate of patients with perioperative complications | 1 month after the surgery
  The perioperative complication includes death, wound infection, hemorrhage, infection, pleural effusion, pneumothorax, cardiovascular problem and etc.

CONTACTS AND LOCATIONS:
Overall Officials: Haiquan Chen, Ph.D, Principal Investigator — Shanghai Cancer Center
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
Study Protocol, Inform Consent Form, Clinical Study Report would not be shared after the study begin.

REFERENCES:
- [Derived] Zhang Y, Qian B, Song Q, Ma J, Cao H, Deng C, Wang S, Ye T, Xiang J, Zhang Y, Sun Y, Yan Y, Zheng S, Wu H, Huang Q, Hu H, Li Y, Fu F, Chen H. Phase III Study of Mediastinal Lymph Node Dissection for Ground Glass Opacity-Dominant Lung Adenocarcinoma. J Clin Oncol. 2025 Oct;43(28):3081-3089. doi: 10.1200/JCO-25-00610. Epub 2025 Jul 21. PMID 40690727